CLINICAL TRIAL: NCT04142736
Title: PRone positioN in Patients With spontanEous ventiLation and Acute Hypoxemic respIratory FailurE
Acronym: PRONELIFE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment rate
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Luis Morales, Study Coordinator, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/68-UCI-HUSC
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Failure With Hypoxia; Respiratory Failure Without Hypercapnia
Keywords: Prone position; Acute Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Prone Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone position (Experimental): Patients with acute hypoxemic respiratory failure from any cause
  Interventions: Other: Prone Position
- Supine position (No Intervention): Patients with acute hypoxemic respiratory failure from any cause

INTERVENTIONS:
Other: Prone Position — The best-fitting and most-tolerated oxygen interface will be used in the prone position--this could be different from patient to patient, and different from what is used in the supine position, and could differ between patients but also institutions (i.e., depending on the availability of masks with or without a reservoir bag and with or without the Venturi system, HFNO, CPAP or NIV). The patient will be placed in the prone position for at least 2 hours, which may be prolonged if the patient is comfortable or interrupted if the patient presents any criteria for prone position discontinuation. After the prone position period, the patient will be rotated to the semi-recumbent supine position for at least 2 hours and a maximum of 4 hours. This 2-hour time frame will depend on nursing availability, need for hygiene, complementary explorations, or diet.
  Arms: Prone position

SUMMARY:
The proposed randomized controlled trial aims at comparing the application of the prone position in spontaneously breathing patients with acute hypoxemic respiratory failure from any cause versus standard treatment on the rate of invasive mechanical ventilation or all-cause of mortality. The secondary endpoints will include time to tracheal intubation and effects of awake proning on the oxygenation parameters, dyspnea sensation, complications, and tolerance. Other endpoints are ventilation free-days at 28 days, duration of invasive ventilation, length of ICU and hospital stay, ICU and hospital mortality, and 28, 60, and 90-day mortality.

DETAILED DESCRIPTION:
The investigators intend to recruit acute hypoxemic respiratory failure patients with a respiratory rate of more than 25 breaths per minute, SpO2 < 94% and FiO2 of at least 40% or more by either Venturi facemask, HFNC, or NIV/CPAP and, absence of decompensated respiratory acidosis during two years. Currently, the investigators expect about 35 centers to participate in the trial.

Demographic data and clinical characteristics on screened patients, regardless of enrolment criteria match, will be recorded (registry). The investigators will randomize 650 patients admitted to the participating centers' intensive care units and expect each participating center to randomize at least 25 patients who meet all inclusion criteria.

ELIGIBILITY:
Inclusion criteria

* >18 years
* Acute respiratory failure from any cause
* Admitted to a participating ICU
* Written informed consent

Exclusion criteria

* Presence of any contraindication to prone position (APPENDIX i)
* The patient meets the criteria for intubation (see item 7.2.3)
* Participating in other interventional studies with the same primary outcome
* Receiving comfort care only
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint comprising the rate of tracheal intubation or all-cause of mortality during the first fourteen days of enrolment. | 14 days

SECONDARY OUTCOMES:
Mortality at day 14 | 14 days
  Effect of prone position on mortality
Intubation among survivors at day 24 | 24 days
  Effect of prone position on the rate of intubation
Effects on oxygenation defined by the SpO2 | 4 hours
  Effects of prone position on oxygenation
Days under the oxygen support device | 28 days
  Days under the oxygen support device (HFNC, NIV, non-rebreather mask, Venturi mask) The VAS is a straight horizontal line of fixed length. The ends are defined as the extreme limits of the parameter to be measured (symptom,pain,health) orientated from the left (worst) to the right (best).
Dyspnea | 4 hours
  Effects of prone position on dyspnea, defined according modified Borg dyspnea scale.
  This is a scale rates the difficulty of breathing. It starts at number 0 where dyspnea is causing no difficulty at all and progresses through to number 10 where dyspnea is maximal.
Time to tracheal intubation | 14 days
  Effects of prone position on timing for tracheal intubation
Rate of complications related to prone position | 4 hours
  Effects of prone position on adverse effects such Oxygen desaturations (SpO2 <90%)
  * Episodes of hemodynamic instability (BPsys < 90mmHg or BPsys drop > 10mmHg if BPsys < 90 before the maneuver)
  * Need of orotracheal intubation
  * Cardiac arrest
  * Displacement of the non-invasive respiratory support device
  * Removal of central venous line, if documented
  * Displacement of an arterial line, if documented
  * Displacement of a urinary catheter, if documented
Respiratory rate | 4 hours
  Effects of prone position of respiratory rate
Duration of invasive mechanical ventilation | 90 days
  Duration of invasive mechanical ventilation in those patients who required intubation
Ventilation-free days (VFD) at 28 days from ICU admission, | 28 days
  Ventilation-free days (VFD) at 28 days from ICU admission, defined as the number of days alive and free from IMV during the first 28 days from start of IMV
ICU-free days and hospital-free days | 90 days
  ICU-free days and hospital-free days at day 90
Mortality | 28 and 90 days
  Mortality at day 28 and day 90

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Artigas, MD, PhD, Principal Investigator — I3PT Institut d'Investigació i Innovació Parc Taulí
Locations (1):
- I3PT Institut d'Investigació i Innovació Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access request will be reviewed by an External Independent Review Panel. Requestors will be required to signed a Data Access Agreement

REFERENCES:
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Scaravilli V, Grasselli G, Castagna L, Zanella A, Isgro S, Lucchini A, Patroniti N, Bellani G, Pesenti A. Prone positioning improves oxygenation in spontaneously breathing nonintubated patients with hypoxemic acute respiratory failure: A retrospective study. J Crit Care. 2015 Dec;30(6):1390-4. doi: 10.1016/j.jcrc.2015.07.008. Epub 2015 Jul 16. PMID 26271685
- [Background] Riera J, Perez P, Cortes J, Roca O, Masclans JR, Rello J. Effect of high-flow nasal cannula and body position on end-expiratory lung volume: a cohort study using electrical impedance tomography. Respir Care. 2013 Apr;58(4):589-96. doi: 10.4187/respcare.02086. PMID 23050520
- [Derived] Morales-Quinteros L, Schultz MJ, Serpa-Neto A, Antonelli M, Grieco DL, Roca O, Juffermans NP, de Haro C, de Mendoza D, Blanch L, Camprubi-Rimblas M, Goma G, Artigas-Raventos A; PRONELIFE collaborative group. Awake prone positioning in nonintubated spontaneous breathing ICU patients with acute hypoxemic respiratory failure (PRONELIFE)-protocol for a randomized clinical trial. Trials. 2022 Jan 10;23(1):30. doi: 10.1186/s13063-021-05991-2. PMID 35012606